CLINICAL TRIAL: NCT02756416
Title: Perfusion MRI in Reversible Cerebral Vasoconstriction Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15085
Record Dates: First submitted 2016-03-02; First posted 2016-04-29 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Reversible Cerebral Vasoconstriction Syndrome
Keywords: Reversible Cerebral Vasoconstriction Syndrome (RCVS); Arterial spin labeling (ASL) MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASL MRI and MRA (Experimental): All participants will undergo ASL-MRI and MRA at three points; baseline, month 1, and month 3.
  Interventions: Device: MRI brain; Device: ASL-MRI brain; Device: MRA brain

INTERVENTIONS:
Device: MRI brain — Standard MRI brain will be performed on each participant to look at brain structure and exclude complications of RCVS (if any).
Device: ASL-MRI brain — ASL-MRI is a non-contrast scan used to measure cortical cerebral blood flow (CBF) in areas supplied by major arteries (Circle of Willis).
Device: MRA brain — MR angiography scan looks at blood vessels structure. We expect to see constriction (narrowing) of the major arteries in RCVS cases.

SUMMARY:
This study aims to quantify perfusion, assess arterial vasoconstriction, and confirm reversibility using 3T ASL-MRI and MRA in 10 patients with suspected RCVS. Acquiring these data at multiple time points during RCVS progression, the investigators will assess the relationship between vasoconstriction and downstream perfusion and determine the role of these imaging techniques in early and accurate diagnosis of RCVS. The investigators also aim to investigate whether early imaging abnormalities can predict RCVS complications and clinical outcomes.

DETAILED DESCRIPTION:
Reversible Cerebral Vasoconstriction Syndrome (RCVS) is a group of conditions characterised by prolonged but reversible multifocal narrowing of the cerebral arteries. It presents typically as acute severe headache, usually recurrent and thunderclap in character, with or without additional symptoms and signs. Adverse complications associated with RCVS can be devastating especially if not recognised early; depending on the degree of vasoconstriction, RCVS may be associated with cortical subarachnoid haemorrhage (in approximately 34% of patients), ischaemic infarction (6-39% of patients), or concomitant posterior reversible encephalopathy syndrome (PRES, 9-38% of patients). RCVS may also present as parenchymal brain haemorrhage in 20% of cases. The data on complications rate highlight the uncertainty about the condition and indicate need for more research to better characterise the evolution of the pathology; hence need for this study as it is prospective and longitudinal.

The hallmark of RCVS is vasoconstriction seen on vascular imaging scans and typically reverses within 3 months. Prevalence of radiological vasoconstriction seen on magnetic resonance angiography (MRA) in RCVS is reported to be between 60-90% and typically appears as diffuse segmental constriction of large and medium sized vessels lasting 4-12 weeks. The main advantage of MRA is that it can be performed without the use of a radioactive tracer, thus providing a safe method for repeat observations of vascular pathology. Imaging is often negative in first 4-5 days following the onset of headache; The mean time to detect abnormality on vascular imaging has been reported as 8 days after headache onset. RCVS symptoms usually resolves by 1 month after presentation, however the adverse complications associated with RCVS may have lasting consequences as described above. Magnetic resonance imaging (MRI) is an excellent tool for characterising brain changes during the progression and resolution of RCVS. Standard structural images can identify complications of RCVS, such as bleeding, ischaemia, and PRES.

Finally, Arterial Spin Labeling (ASL) MRI can be used to non-invasively quantify perfusion of brain tissue, providing a measure of the impact of upstream arterial vasoconstriction on local cortical regions.

Cortical perfusion has not yet been extensively studied in RCVS; at time of writing, only two case reports have been published. Rosenbloom and Singhal reported a case of RCVS induced by carotid endarterectomy following a frontal lobe ischaemic stroke. Perfusion MRI showed unilateral hypo-perfusion, mainly affecting internal watershed areas with superficial cortical regions being relatively spared. In a second study, ASL-MRI was performed on a 50-year-old man with RCVS who presented with severe recurrent headaches and neurological deficits (localising to the right hemisphere). ASL-MRI demonstrated significant hypo-perfusion in the right parieto-occipital lobe, but no infarct was seen on diffusion imaging. At 12 weeks, there was complete resolution of cerebral vasoconstriction on angiography and normal perfusion findings on ASL-MRI.

These case studies suggest that perfusion MRI can offer an additional tool to confirm and understand RCVS. ASL-MRI is a non-invasive, radiation and contrast-free technique that can be performed at multiple time points to monitor changes in perfusion over the time period of RCVS resolution and assess response to potential therapeutics.

One of the disadvantages of ASL-MRI is a low signal to noise ratio, this can be addressed by using high-field MRI at 3 Tesla (3T). In addition, 3T MRI can provide very good spatial resolution. The University of Nottingham represents one of the leading international research centres with experience in using high and ultra-high field MRI for investigating different neurological diseases such as multiple sclerosis and brain tumours with excellent results. Applying advanced non-invasive MRI techniques in this study will be a significant advantage as we investigate RCVS, understand the pathophysiology, and assess brain perfusion in multiple time points.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18-60 years old
* Able to give informed written consent
* Clinical presentation suggestive of RCVS
* Able to understand the requirements of the study, including anonymous publication, and agree to co-operate with the study procedures

Exclusion Criteria:

* Evidence of brain haemorrhage or significant brain pathology on Computed Tomography (CT) scan performed as standard National Health Service (NHS) care
* Any history of significant cerebrovascular disease
* Pregnancy or breastfeeding
* MRI contraindications (e.g. metal implants or pacemaker) as indicated on the MRI Safety Screening Questionnaire
* Significant claustrophobia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change in cortical cerebral blood flow (CBF) measured in ml/100g/min using ASL-MRI. | Baseline, month 1, and month 3
  The process includes detailed imaging analysis.
Change in Circle of Willis arteries and major branches structure, this will be assessed by MRA and examined by a neuro-radiologist. | Baseline, month 1, and month 3
  Correlation between vascular changes and perfusion levels will be measured.

SECONDARY OUTCOMES:
RCVS complications, such as ischaemia, bleeding, and posterior reversible encephalopathy syndrome, will be assessed using standard MRI brain sequences. | Baseline, month 1, and month 3
  Correlation between occurrence of these complications and perfusion levels will be measured.
Headache characteristics; participants will be questioned about their headache using a questionnaire as part of the case report form. | Baseline, month 1, and month 3
  Correlation between headache characteristics and perfusion levels will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Neurology, Division of Clinical Neuroscience, University of Nottingham, UK, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Calabrese LH, Dodick DW, Schwedt TJ, Singhal AB. Narrative review: reversible cerebral vasoconstriction syndromes. Ann Intern Med. 2007 Jan 2;146(1):34-44. doi: 10.7326/0003-4819-146-1-200701020-00007. PMID 17200220
- [Background] Ducros A, Boukobza M, Porcher R, Sarov M, Valade D, Bousser MG. The clinical and radiological spectrum of reversible cerebral vasoconstriction syndrome. A prospective series of 67 patients. Brain. 2007 Dec;130(Pt 12):3091-101. doi: 10.1093/brain/awm256. Epub 2007 Nov 19. PMID 18025032
- [Background] Miller TR, Shivashankar R, Mossa-Basha M, Gandhi D. Reversible Cerebral Vasoconstriction Syndrome, Part 1: Epidemiology, Pathogenesis, and Clinical Course. AJNR Am J Neuroradiol. 2015 Aug;36(8):1392-9. doi: 10.3174/ajnr.A4214. Epub 2015 Jan 15. PMID 25593203
- [Background] Bernard KR, Rivera M. Reversible Cerebral Vasoconstriction Syndrome. J Emerg Med. 2015 Jul;49(1):26-31. doi: 10.1016/j.jemermed.2015.01.012. Epub 2015 Apr 7. PMID 25858343
- [Background] Sattar A, Manousakis G, Jensen MB. Systematic review of reversible cerebral vasoconstriction syndrome. Expert Rev Cardiovasc Ther. 2010 Oct;8(10):1417-21. doi: 10.1586/erc.10.124. PMID 20936928
- [Background] Lee R, Ramadan H, Bamford J. Reversible cerebral vasoconstriction syndrome. J R Coll Physicians Edinb. 2013;43(3):225-8. doi: 10.4997/JRCPE.2013.307. PMID 24087801
- [Background] Calic Z, Cappelen-Smith C, Zagami AS. Reversible cerebral vasoconstriction syndrome. Intern Med J. 2015 Jun;45(6):599-608. doi: 10.1111/imj.12669. PMID 25511128
- [Background] Mortimer AM, Bradley MD, Stoodley NG, Renowden SA. Thunderclap headache: diagnostic considerations and neuroimaging features. Clin Radiol. 2013 Mar;68(3):e101-13. doi: 10.1016/j.crad.2012.08.032. Epub 2012 Dec 11. PMID 23245274
- [Background] Dilli E. Thunderclap headache. Curr Neurol Neurosci Rep. 2014 Apr;14(4):437. doi: 10.1007/s11910-014-0437-9. PMID 24643327
- [Background] Miller TR, Shivashankar R, Mossa-Basha M, Gandhi D. Reversible Cerebral Vasoconstriction Syndrome, Part 2: Diagnostic Work-Up, Imaging Evaluation, and Differential Diagnosis. AJNR Am J Neuroradiol. 2015 Sep;36(9):1580-8. doi: 10.3174/ajnr.A4215. Epub 2015 Jan 22. PMID 25614476
- [Background] Rosenbloom MH, Singhal AB. CT angiography and diffusion-perfusion MR imaging in a patient with ipsilateral reversible cerebral vasoconstriction after carotid endarterectomy. AJNR Am J Neuroradiol. 2007 May;28(5):920-2. PMID 17494670
- [Background] Komatsu T, Kimura T, Yagishita A, Takahashi K, Koide R. A case of reversible cerebral vasoconstriction syndrome presenting with recurrent neurological deficits: Evaluation using noninvasive arterial spin labeling MRI. Clin Neurol Neurosurg. 2014 Nov;126:96-8. doi: 10.1016/j.clineuro.2014.08.023. Epub 2014 Aug 30. No abstract available. PMID 25238101